CLINICAL TRIAL: NCT05812287
Title: Exploring the Difference Between Gastric Cardia Cancer and Non-cardia Gastric Cancer Based on Multiomics
Status: Not yet recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023SDU-QILU-2
Record Dates: First submitted 2023-04-02; First posted 2023-04-13 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-03

CONDITIONS: Stomach Neoplasm
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: The case group includes high-grade intraepithelial neoplasia of the stomach, early gastric cancer, and advanced gastric cancer. According to the anatomical location of the tumors, they were divided into two groups: gastric cardia cancer and non-cardia gastric cancer.
  Interventions: Other: Detection of biological samples based on multi-omics analysis
- Control: Pathological findings in the control group showed no malignant changes in the stomach, including normal gastric mucosa, superficial gastritis, non atrophic gastritis, and gastric polyps, etc.
  Interventions: Other: Detection of biological samples based on multi-omics analysis

INTERVENTIONS:
Other: Detection of biological samples based on multi-omics analysis — In this study, we combined microbiological (16SrRNA) and metabolomic mass spectrometry to study the changes in microbial populations and metabolic profiles of various samples such as feces, serum, and saliva, and screen key differential markers.

SUMMARY:
This is an observational study with a case control design. This study included patients with gastric cancer confirmed by pathological diagnosis of gastric tissue, and matched the control population according to age, gender, etc. In this study, researchers collected clinical information and multiple biological samples such as saliva, serum, and feces from the study subjects. We combined 16S rRNA sequencing and metabolomics to explore the differences in microbial and metabolic characteristics between gastric cardia cancer and non-cardia gastric cancer for early screening of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Study population signing informed consent form
* Age: 18-75 years old
* The study population must underwent endoscopic examination and was confirmed by pathological diagnosis as gastric cancer: including high-level intraepithelial neoplasia, early gastric cancer, and advanced gastric cancer.

Exclusion Criteria:

* Those who have undergone gastrointestinal surgery within the past 1 year; Patients who have undergone neoadjuvant chemotherapy and have developed tumors in the residual stomach after previous partial gastrectomy.
* Those who have used proton pump inhibitors, antibiotics, probiotics, and prebiotics daily within the past month, and those who have recently received hormone therapy.
* People with infectious diseases and other digestive system diseases that interfere with the experimental results, such as inflammatory bowel disease, irritable bowel syndrome, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case:
  The population in the case group signed an informed consent form, aged between 18 and 75 years. All subjects underwent endoscopic examination and were confirmed by pathological diagnosis as gastric cancer, including high-grade intraepithelial neoplasia, early gastric cancer, and advanced gastric cancer.
  Control:
  The age and gender of the study subjects in the control group were matched to the study population in the case group. The pathological results of the stomach of all subjects showed no malignant changes, including normal gastric mucosa, superficial gastritis, non atrophic gastritis, and gastric polyps, etc.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Early gastric cancer detection rate | 36 months
  This study combines 16SrRNA sequencing and metabolomics to explore the differences in microbiota and metabolites between tumor cohorts and healthy controls, and to assist in screening for early gastric cancer.